CLINICAL TRIAL: NCT02099903
Title: Transcatheter Renal Denervation in Patients With Systolic Heart Failure Due to Chagas' Disease - a Safety and Efficacy Study.
Brief Title: Renal Denervation in Patients With Heart Failure Secondary to Chagas Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: InCor Heart Institute (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Pedro A. Lemos, Professor of Medicine, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18400613.1.0000.0068
Record Dates: First submitted 2014-03-19; First posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Heart Failure; Heart Failure, Systolic; Chagas Disease; Chagas Cardiomyopathy
Keywords: Heart Failure; Heart Failure, Systolic; Chagas Disease; Chagas Cardiomyopathy; Renal Denervation; Irrigated Radiofrequency Catheter
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Chagas Disease; Chagas Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical therapy for heart failure (No Intervention): Standard optimized medical therapy for heart failure.
- Renal denervation + medical therapy. (Experimental): Transcatheter Renal Denervation with irrigated radiofrequency catheter + standard medical therapy.
  Interventions: Device: transcatheter renal denervation

INTERVENTIONS:
Device: transcatheter renal denervation — Renal sympathetic denervation with an irrigated radiofrequency catheter.
  Other Names: Celsius Thermocool (Biosense Webster, California, USA)
  Arms: Renal denervation + medical therapy.

SUMMARY:
It is a randomized prospective controlled study of transcatheter renal denervation in patients with systolic heart failure secondary to Chagas' disease. The purpose of the study is to evaluate the safety and effectiveness of renal denervation in patients with Chagas heart disease, due to reduction in renal and systemic sympathetic activity.

DETAILED DESCRIPTION:
The activation of the sympathetic nervous system is one of the main mechanisms involved in heart failure pathophysiology, as well as activation of the renin-angiotensin-aldosterone system. These compensatory mechanisms are initially beneficial, in order to restore adequate cardiac output. Their long-term activation, nevertheless, leads to several deleterious effects on cardiovascular system, such as direct myocite lesion, cardiac hypertrophy, myocardial ischemia, oxidative stress, cardiac arrhythmias and myocite apoptosis, among others.

It has been widely demonstrated that modulation of sympathetic nervous system is an important therapeutic target for the treatment of systolic heart failure. Beta-blocker and ACE inhibitors therapies are the main stem of heart failure treatment and have demonstrated reduction in morbidity and mortality of this condition. Despite optimized medical treatment, heart failure carries a poor prognosis.

Surgical sympathectomy has been used decades ago for the treatment of malignant hypertension and showed marked reduction in arterial pressure. However, these procedures were very aggressive and lead to long hospitalization and recovery periods, as well as several limiting adverse effects. Recently, transcatheter renal denervation has evolved as a promising and less invasive technique, which allows destruction of renal nerves located on the adventitia of the renal arteries. The ablation procedure is performed by delivery of radiofrequency energy from the tip of a catheter positioned into the renal arteries, through standard femoral artery catheterization, a less morbid and safer approach.

Renal denervation has been tested mainly in patients with resistant hypertension, among other indications, with promising results. The pathophysiological basis for this treatment in hypertension, as well as heart failure, stands on the participation of renal afferent and efferent nerves on the maintenance of elevated systemic vascular resistance. Activation of efferent nerves leads to excretion o renin, aldosterone, angiotensin II, elevated norepinephrine levels and consequent retention of salt and water and reduction of renal blood flow. This mechanism and also afferent renal nerves activation contributes to the elevation of sympathetic tonus on the central nervous system.

In animal models of heart failure, renal denervation demonstrated improvement on renal and cardiac function. Initial clinical studies suggest that this intervention is safe and potentially effective on the treatment of heart failure in humans. Chagas heart disease is a prevalent cause of heart failure in Brazil and shares several pathophysiological aspects described for other causes of heart failure. Our aim is to evaluate the safety and effectiveness of renal denervation in systolic heart failure due to Chagas Heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 to ≤ 70 years of age with chronic systolic heart failure, Chagas disease etiology.
2. Two positive serology results for Chagas by two distinct methods.
3. NYHA (New York Heart Association) class II or III.
4. Patients treated with maximum tolerated doses of standard pharmacotherapy for heart failure.
5. LVEF (Left Ventricular Ejection Fraction) ≤ 40% (Simpson Method).

Exclusion Criteria:

1. Patients with NYHA class I or IV.
2. Sustained ventricular tachycardia (>30 sec) or with hemodynamic compromise.
3. Presence of permanent pacemaker or implantable defibrillator.
4. Systolic blood pressure < 90 mmHg.
5. Heart beat < 60 bpm at rest.
6. Advanced renal insufficiency (estimated glomerular filtration rate (GFR) < 30 ml/min/1.73 square meters).
7. Patients with planned cardiac surgery or percutaneous revascularization.
8. Other reasons which would preclude the patient from participating in the study (comorbidities, life expectancy less than 1 year).
9. Unsuitable anatomy of renal arteries, renal stenosis or previous treatment with balloon or stent.
10. Refusal of the patient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Composite: death, myocardial infarction, cerebrovascular event, need of intervention on renal arteries and renal function impairment (decrease in estimated GFR > 30% from baseline). | 30 days.

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) by echocardiography. | 9 months.
New York Heart Association (NYHA) functional class. | 9 months.
6-minute walk test | 9 months.
Peak Oxygen consumption (VO2) by ergoespirometry. | 9 months.

OTHER OUTCOMES:
Change in serum B-type natriuretic peptide (BNP). | 9 months.
Quality of life assessed by Minnesota and EuroQOL five dimensions (EQ-5D)questionnaires. | 9 months.
Peripheral sympathetic activity measured by microneurography. | 9 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute - InCor. University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil